CLINICAL TRIAL: NCT01320761
Title: A Study to Assess Injection Comfort of Two Formulations of ATX-101 (Sodium Deoxycholate Injection) Following Subcutaneous Administration in the Submental Area
Brief Title: A Study to Assess Injection Comfort of Two Formulations of ATX-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Daniel R. Lee, M.S., Director, Clinical Affairs, Kythera Biopharmaceuticals, Inc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATX-101-10-19
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Healthy
Keywords: Formulation Comparison

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1A (Experimental): Left side injected first:
  Left submental - ATX-101-BA Right submental - ATX-101-BA-free
  Interventions: Drug: ATX-101-BA-free; Drug: ATX-101-BA
- Group 1B (Experimental): Right side injected first:
  Left submental - ATX-101-BA Right submental - ATX-101-BA-free
  Interventions: Drug: ATX-101-BA-free; Drug: ATX-101-BA
- Group 2A (Experimental): Left side injected first:
  Left submental - ATX-101-BA-free Right submental - ATX-101-BA
  Interventions: Drug: ATX-101-BA-free; Drug: ATX-101-BA
- Group 2B (Experimental): Right side injected first:
  Left submental - ATX-101-BA-free Right submental - ATX-101-BA
  Interventions: Drug: ATX-101-BA-free; Drug: ATX-101-BA

INTERVENTIONS:
Drug: ATX-101-BA-free — ATX-101-BA-free
Drug: ATX-101-BA — ATX-101-BA

SUMMARY:
To assess the safety and injection comfort of ATX-101-BA versus ATX-101-BA-free immediately following injection and at regular intervals up to 24-hours post-injection following subcutaneous administration into the submental area.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of submental fat graded by the investigator as 2, 3, or 4 using the CR-SMFRS (Appendix B).
2. Sufficient and symmetrical submental fat such that the protocol-specified number of injections can be safely administered on both the right and left side.
3. No difference in perception or sensitivity (pain or otherwise) between left and right sides of the submental area.
4. Abstinence from alcohol for at least 6 hours prior to both the Baseline and 24-hour visits.
5. Males or nonpregnant, nonlactating females who are aged 18 to 65 years, inclusive, on Baseline date.
6. Females of child-bearing potential must have a negative urine human chorionic gonadotropin (hCG) test result from a sample obtained during the screening period. Females of childbearing potential must agree to practice adequate contraception, in the judgment of the investigator, during the course of the trial (including post-screening).
7. The subject is expected to comply with and understand the visit schedule and all of the protocol-specified tests and procedures.
8. The subject is medically able to undergo the administration of study material as determined by clinical and laboratory evaluations obtained within 14 days before dosing with study material for which the investigator identifies no clinically significant abnormality.
9. Signed informed consent obtained before any study-specific procedure is conducted.

Exclusion Criteria:

1. History of any intervention (e.g., liposuction) or trauma associated with the chin or neck areas, which in the judgment of the investigator, may affect subject safety or other evaluations of treatment.
2. Evidence of any cause of enlargement in the submental area (e.g., thyroid enlargement, cervical adenopathy) other than localized submental fat.
3. Any medical condition (e.g., respiratory, cardiovascular, hepatic, neurological disease, uncontrolled hypertension, thyroid dysfunction), that would interfere with the assessment of safety in this trial or would compromise the ability of the subject to undergo study procedures or to give informed consent.
4. Any cognitive impairment that, in the Investigator's opinion, would preclude study participation or compliance with protocol-specified procedures.
5. Treatment with analgesics or other agents that could affect the pain response, including but not limited to acetaminophen or ibuprofen taken within 1 day prior to Baseline; additionally, narcotic analgesics, tranquilizers, hypnotics, sedatives, or opiates within 7 days prior to Baseline.
6. Treatment of the chin or SMF with injectable steroids within 90 days prior to Baseline.
7. Participation in a pain study within 6 months prior to Baseline.
8. History of chronic pain and/or a history of chronic analgesic or tranquilizer use within 90 days prior to Baseline.
9. Any anticipated need for agents with anticoagulative effects (e.g., aspirin, ibuprofen, warfarin, heparin) during the course of the trial.
10. Treatment with oral anticoagulants (e.g., aspirin, warfarin) within 10 days prior to Baseline.
11. Treatment with topical agents to the submental or neck area, including but not limited to creams or ointments used to treat dermatologic conditions (e.g., steroids, capsaicin, retinoids, fluorouracil) within 7 days prior to Baseline.
12. Treatment with radio frequency, laser procedures, chemical peel, or dermal fillers in the neck or chin area within 12 months before dosing or botulinum toxin injections within 6 months prior to Baseline.
13. Previous enrollment into this trial or treatment with ATX-101 or agents containing deoxycholate.
14. Treatment with an investigational agent within 28 days prior to Baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)

PRIMARY OUTCOMES:
Comfort measure | up to 24 hours after treatment
  The primary measure of comfort is the pain comparison scale between ATX-101-BA and ATX-101-BA-free at the time of injection using the pain comparison scale and the VAS pain rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Walker, M.D., Study Director — Kythera Biopharmaceuticals, Inc
Locations (2):
- United States (2):
  - Joel Schlessinger, M.D., Omaha, Nebraska
  - Jeffrey M. Adelglass, M.D., Plano, Texas